CLINICAL TRIAL: NCT05086081
Title: Replication of the ISAR-REACT 5 Antiplatelet Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-ISAR-REACT5
Record Dates: First submitted 2021-09-20; First posted 2021-10-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prasugrel: Reference group
  Interventions: Drug: Prasugrel 10mg
- Ticagrelor: Exposure group
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Any ticagrelor dispensing claim is used as the exposure group
  Groups: Ticagrelor
Drug: Prasugrel 10mg — Any prasugrel dispensing claim is used as the reference group
  Groups: Prasugrel

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Criteria:

Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Inclusion Criteria:

* Hospitalization for unstable angina or acute MI AND age >= 18 years Days [ACS admission]
* STEMI OR NSTEMI/unstable angina (during admission) + 1 of the following

  * >= 60 years old Days [ACS]
  * >= 3 risk factors for coronary artery disease
  * Diabetes mellitus
  * Chronic renal disease
  * Carotid stenosis >= 50% or cerebral revascularization
  * Peripheral artery disease Days [-365, ACS]
  * Aspirin use
  * Angina Days [-7, ACS]
  * Prior MI or CABG any time prior

Exclusion Criteria:

* Acute complication PCI Days [-30, ACS admission]
* History of any stroke or TIA Days [all available data, 0]
* Intracranial neoplasm, intracranial AVM, intracranial neoplasm Days [-180, 0]
* Active bleeding Days [-180, 0]
* Platelet count < 100.000/uL Days [-180, 0]
* Anemia (hemoglobin < 10 g/dL) Days [-180, 0]
* Chronic renal insufficiency requiring dialysis Days [-180, 0]
* Moderate to severe hepatic dysfunction Days [-180, 0]
* Increased risk of bradycardia events Days [-180, 0]
* Life expectancy, 1 year Days [-180, 0]
* Pregnancy Days [-180, 0]
* Concomitant therapy CYP3A inhibitors, CYP3A substrates, or strong CYP3A inducers Days [-14, 0]

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, retrospective cohort study design comparing ticagrelor 90 mg twice daily to prasugrel 10 mg daily. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of ticagrelor or prasugrel (index date). We will restrict the analyses to patients with an acute coronary syndrome, with or without ST-segment elevation, who were scheduled to undergo coronary angiography.
Sampling Method: Probability Sample
Enrollment: 28389 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite of death, myocardial infarction, or stroke at 1 year after randomization | Through study completion or censoring, up to 12 months
  Claims-based algorithm: Relative hazard of composite of death, myocardial infarction, or stroke at 1 year after randomization

SECONDARY OUTCOMES:
Relative hazard of hospital admission for MI, hospital admission for stroke, or death | Through study completion or censoring, up to 12 months
  Claims-based algorithm: Relative hazard of hospital admission for MI, hospital admission for stroke, or death
Relative hazard of major bleeding | Through study completion or censoring, up to 12 months
  Claims-based algorithm: relative hazard of major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT05086081/Prot_000.pdf